CLINICAL TRIAL: NCT02452736
Title: CHINA RESOLUTE INTEGRITY STUDY Acute Safety, Deliverability and Efficacy of the Medtronic Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System in the Treatment of Suitable Patients According to Indication for Use --A Prospective, Multi-center, Single Arm, Non-randomized Study
Brief Title: Acute Safety, Deliverability and Efficacy of the Medtronic Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System in the Treatment of Suitable Patients According to Indication for Use (CHINA RESOLUTE INTEGRITY STUDY)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-Resolute Integrity China
Record Dates: First submitted 2015-05-01; First posted 2015-05-25 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Ischemic Heart Disease; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Ischemia; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System (Experimental): This is a Single arm, Non-randomized Study. All patients meet the eligibility criteria and sign the informed consent form will participate in this study.
  Interventions: Device: Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System

INTERVENTIONS:
Device: Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System

SUMMARY:
The purpose of this study is to conduct a prospective, multi-center, single arm, non-randomized evaluation of acute outcomes in Chinese subjects, including those eligible for percutaneous transluminal coronary angioplasty (PTCA) with a reference vessel diameter of 2.25 mm to 4.0 mm, with the Medtronic Resolute Integrity™ Zotarolimus-Eluting Coronary Stent System.

DETAILED DESCRIPTION:
This is a Pre-market, Prospective, Multi-center, Single arm, Non-randomized Study.

The objective of this study is to:

* To assess the deliverability of the Resolute Integrity Stent for suitable patients according to Indication for Use with a reference vessel diameter (RVD) of 2.25 mm to 4.0 mm in 200 evaluable patients
* To assess the in-hospital Major Adverse Cardiac Event (MACE) rate
* To collect data on resource utilization in the catheterization lab. At least 200 evaluable patients from about 15 study centers in China who meet the eligibility criteria and sign the informed consent form will participate in this study.

The expected time of participation in the study for each subject is from informed consent sign-off up to hospital discharge.

An angiographic core laboratory and a Clinical Events Committee (CEC) will be utilized. Adjudication of pre-specified clinical endpoint events will be done by an independent Clinical Events Committee. An angiographic core laboratory will review all baseline, procedural, and clinical event angiograms for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is older than or equal to 18 years
2. The patient is an acceptable candidate for treatment with a drug-eluting stent in accordance with the applicable guidelines on percutaneous coronary interventions, the Instructions for Use of the Resolute Integrity stent
3. The patient or legal representative has been informed of the nature of the trial and has consented to participate and authorized the collection and release of his/her medical information by signing a Patient Informed Consent Form
4. Intention to implant at least one Resolute Integrity stent during percutaneous coronary intervention (PCI)
5. Patient agrees to have all study procedures performed, and is willing to comply with all protocol-required evaluations

Exclusion Criteria:

1. Known hypersensitivity or contraindication to aspirin, heparin and bivalirudin, clopidogrel and ticlopidine, cobalt, nickel, chromium, molybdenum, polymer coatings (e.g. BioLinx) or a sensitivity to contrast media, which cannot be adequately pre-medicated
2. History of an allergic reaction or significant sensitivity to drugs such as zotarolimus, rapamycin, tacrolimus, everolimus, or any other analogue or derivative
3. A woman who is pregnant, planning to be pregnant or lactating
4. Currently participating in another trial
5. Situation that will prevent dual anti-platelet therapy to be maintained throughout the peri-surgical period
6. Previous enrollment in the China Resolute Integrity Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Device Specific Procedural Success | Participants will be followed for the duration of hospital stay, an expected average of 5 days.
  Defined as device success (the attainment of less than 50% residual stenosis of the target lesion using only the study device) and no in-hospital MACE (composite of death, myocardial infarction, emergent coronary bypass surgery, or clinically-driven repeat target lesion revascularization).

SECONDARY OUTCOMES:
Delivery Success | Participants will be followed at the end of index procedure, an expected average of 3 days.
  Defined as complete passage of the Resolute Integrity stent across the target lesion with full expansion of the stent to the desired diameter at the desired location.
Device Success | Participants will be followed at the end of index procedure, an expected average of 3 days.
  defined as the attainment of less than 50% residual stenosis of the target lesion using only the Resolute Integrity stent.
Lesion Success | Participants will be followed at the end of index procedure, an expected average of 3 days.
  Defined as the attainment of less than 50% residual stenosis by any percutaneous method.
Procedure Success | Participants will be followed for the duration of hospital stay, an expected average of 5 days.
  Defined as the attainment of less than 50% residual stenosis by any percutaneous method and no in-hospital MACE.
In-hospital Major Adverse Cardiac Events (MACE) | Participants will be followed for the duration of hospital stay, an expected average of 5 days.
  Defined as the composite of as in-hospital death, myocardial infarction (Q-wave and non Q-wave), emergent coronary bypass surgery, or repeat target lesion revascularization (TLR; clinically driven/clinically indicated) by percutaneous or surgical method.
In-hospital Target Lesion Failure (TLF) | Participants will be followed for the duration of hospital stay, an expected average of 5 days.
  Defined as the composite of cardiac death, myocardial infarction (not clearly attributable to a non-target vessel) or target lesion revascularization (TLR; clinically indicated).
Procedure time (min) | Participants will be followed at the end of index procedure, an expected average of 3 days.
  Resource Utilization
Contrast volume used (ml) | Participants will be followed at the end of index procedure, an expected average of 3 days.
  Resource Utilization
Usage of guiding catheters | Participants will be followed at the end of index procedure, an expected average of 3 days.
  Resource Utilization
Usage of guide wires | Participants will be followed at the end of index procedure, an expected average of 3 days.
  Resource Utilization
Usage of angioplasty balloons | Participants will be followed at the end of index procedure, an expected average of 3 days.
  Resource Utilization

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Nanjing First Hospital, Nanjing, Jiangsu